CLINICAL TRIAL: NCT02433093
Title: A Single-Center, Randomized, Investigator/Participant-Blind, Placebo-Controlled, Multiple-Ascending Dose, Semi-Sequential Adaptive Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Basimglurant Following Oral Administration in Healthy Subjects and in Patients With Major Depressive Disorder
Brief Title: A Study of the Safety, Tolerability, and Pharmacokinetics of Multiple-Ascending Dose Basimglurant in Healthy Subjects and in Patients With Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: NP29583
Record Dates: First submitted 2015-04-29; First posted 2015-05-04 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Major Depressive Disorder, Healthy Volunteer
MeSH Terms: conditions — Depressive Disorder, Major | interventions — 2-chloro-4-(1-(4-fluorophenyl)-2,5-dimethyl-1H-imidazol-4-ylethynyl)pyridine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (7):
- Basimglurant: Healthy Cohort (1) (Experimental): Healthy participants assigned to basimglurant will receive a 22-day ascending dose regimen. Cohort 1 will receive a prespecified titration scheme; however, adaptive titration schemes may be applied in subsequent cohorts.
  Interventions: Drug: Basimglurant
- Basimglurant: Healthy Cohort (2) (Experimental): Healthy participants assigned to basimglurant will receive a 22-day ascending dose regimen. The dosing scheme for Cohort 2 will be selected in accordance with decision criteria on the basis of the incidence of severe AEs in Cohort 1.
  Interventions: Drug: Basimglurant
- Basimglurant: Healthy Cohort (3) (Experimental): Healthy participants assigned to basimglurant will receive a 22-day ascending dose regimen. The dosing scheme for Cohort 3 will be selected in accordance with decision criteria on the basis of the incidence of severe AEs in preceding Cohorts 1 and 2.
  Interventions: Drug: Basimglurant
- Basimglurant: Healthy Cohort (4) (Experimental): Healthy participants assigned to basimglurant will receive a 22-day ascending dose regimen. The dosing scheme for Cohort 4 will be selected in accordance with decision criteria on the basis of the incidence of severe AEs in preceding Cohorts 1, 2, and 3.
  Interventions: Drug: Basimglurant
- Basimglurant: MDD Cohort (5) (Experimental): Participants with MDD assigned to basimglurant will receive a 22-day ascending dose regimen. The dosing scheme for Cohort 5 may differ from those previously evaluated; however, the titration steps and the highest dose tested will remain equal to or lower than the doses tested in Cohorts 1 to 4.
  Interventions: Drug: Basimglurant
- Placebo: Healthy Cohorts (1 to 4) (Placebo Comparator): Healthy participants will receive a 22-day regimen of matching placebo capsules.
  Interventions: Drug: Placebo
- Placebo: MDD Cohort (5) (Placebo Comparator): Participants with MDD will receive a 22-day regimen of matching placebo capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Basimglurant — Participants will receive once-daily oral basimglurant capsules in a multiple ascending dose regimen. Basimglurant dose will be titrated over 22 days; dose escalations will be separated by at least 4 days, with the final dose administered for a minimum of 14 days. The minimum starting dose will be 1.5 mg, which can be titrated up to a maximum dose of 4.0 mg. Intrapatient dose increments will not exceed 1.0 mg every 4 days.
  Arms: Basimglurant: Healthy Cohort (1); Basimglurant: Healthy Cohort (2); Basimglurant: Healthy Cohort (3); Basimglurant: Healthy Cohort (4); Basimglurant: MDD Cohort (5)
Drug: Placebo — Participants will receive 22 days of once-daily oral matching placebo capsules.
  Arms: Placebo: Healthy Cohorts (1 to 4); Placebo: MDD Cohort (5)

SUMMARY:
The study will assess the safety, tolerability, and pharmacokinetics of basimglurant compared to placebo after multiple ascending oral doses for up to 22 days in healthy subjects and in patients with MDD on stable selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) background therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age, inclusive
* Body weight at least 50 kg
* Healthy male or female subjects (Healthy Cohorts)
* Body mass index (BMI) 18 to 30 kg/m^2, inclusive (Healthy Cohorts)
* Nonsmoker for at least 90 days prior to dosing (Healthy Cohorts)
* Primary diagnosis of MDD without psychotic features (MDD Cohort)
* BMI 18 to 35 kg/m^2, inclusive (MDD Cohort)
* Current partial response to ongoing SSRI or SNRI antidepressant treatment at an adequate dose and for at least 4 weeks (MDD Cohort)
* Clinical Global Impression of Severity (CGI-S) score 3 or greater (MDD Cohort)
* Other regimens stable for at least 8 weeks prior to screening (MDD Cohort)

Exclusion Criteria:

* Pregnant or lactating women
* History of alcohol or substance abuse in the past 6 months
* Hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
* Clinically relevant electrocardiogram (ECG) abnormalities or a personal or family history of congenital long QT syndrome
* Participation in an investigational study within 90 days of screening
* Blood donation over 500 mL within 3 months of screening
* Hypersensitivity to any study medication or excipients
* Psychotic symptoms or comorbid mood disorder
* Significant suicide risk
* Major illness within 1 month before screening, or febrile illness within 1 week (Healthy Cohorts)
* Average alcohol consumption of more than 2 units per day (Healthy Cohorts)
* Multi-drug therapy for depression including antidepressants or adjunctive medications (MDD Cohort)
* Prior use of basimglurant (MDD Cohort)
* Cigarette use of greater than 1 pack per day (MDD Cohort)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events (AEs) | Up to 10 weeks
Safety: Suicidality as assessed using the Columbia Suicide Severity Rating Scale (C-SSRS) | Up to 10 weeks
Safety: Sleep habits as assessed using a participant-recorded sleep diary | Up to 21 days

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum plasma concentration (Cmax) | Post dose on Day 1 and Day 22 (or final dose)
Pharmacokinetics: Area under the plasma concentration-time curve from 0 to 24 hours (AUC0-24) | Post dose on Day 1
Pharmacokinetics: Area under the plasma concentration-time curve over the dosing interval (AUC0-tau) | Post dose on Day 22 (or final dose)
Pharmacokinetics: Time to maximum plasma concentration (Tmax) | Post dose on Day 1 and Day 22 (or final dose)
Pharmacokinetics: Trough plasma concentration (Ctrough) | Post dose on Day 1 and Day 22 (or final dose)
Pharmacokinetics: Apparent terminal elimination half-life (t1/2) | Post dose on Day 22 (or final dose)
Safety: QT interval corrected using the Fridericia method (QTcF) | Up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Garden Grove, California, United States